CLINICAL TRIAL: NCT03300700
Title: Cardiopulmonary Exercise Test in Patient With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nafady, Principal Investigator, Assiut University
Other Study IDs: CETIPWOSA
Record Dates: First submitted 2017-08-29; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea (OSA) can be described as a condition characterized by repetitive obstruction of the upper airway resulting in oxygen desaturation and awakening from sleep, loud snoring, and increased daytime sleepiness . Many studies have shown that a link exists between OSA and cardiovascular disease, chronic heart failure ischemia, hypertension, obesity, and impaired glucose tolerance . A number of factors are likely to play role in development of clinical OSA syndrome (OSAS) ranging from upper airway anatomy to central respiratory control mechanisms. The pathophysiology of OSA is unclear and complex. Several previous studies have explored pulmonary function in the OSAS patients Interestingly, OSAS has been found to be highly correlated with lower airway obstruction, although it is originally defined as an upper airway disease

DETAILED DESCRIPTION:
American Sleep Apnea Association considers exercise as a non-pharmacological treatment modality of sleep disorders . Theoretical reviews and hypotheses on the effects of exercise in OSA have suggested thermoregulatory, metabolic, and biochemical mechanisms although clinical trials on the topic are inadequate .

Cardiopulmonary exercise testing (CPET) is used as a stress test to evaluate cardiac, pulmonary, and muscle function. It has also been used to differentiate whether the etiology of impairment of the ca. rdiopulmonary exercise test is cardiac, pulmonary or muscle dysfunction In otherwise healthy subjects, exercise limitation is due to heart disease. Patients with OSAS are frequently overweight and may exhibit lung function abnormalities related to their weight. These include a decrease in the functional residual capacity (FRC) due mainly to a decrease in the expiratory reserve volume (ERV) and a decrease in compliance of the respiratory system. These functional abnormalities cause an increase in the energy cost of breathing. In addition, increased body mass is associated with greater metabolic energy requirements during muscular exercise, resulting in further ventilatory stress. There are reports demonstrating that there are discriminating measurements during exercise in obesity, including a high O2 cost to perform external work, and upward displacement of the VO2 -WR relationship OSAS patients have daytime hypersomnolence, decreased daily activity and tissue hypoxemia which may further impair muscle function and decrease exercise fitness. Recently, Peppard and Young (2004) found that, independent of body habitus, lack of exercise was associated with increased severity of sleep-disordered breathing measurements during exercise in obesity, including a high O2 cost to perform external work, and upward displacement of the VO2 -WR relationship. OSAS patients have daytime hypersomnolence, decreased daily activity and tissue hypoxemia which may further impair muscle function and decrease exercise fitness. Recently, Peppard and Young (2004) found that, independent of body habitus, lack of exercise was associated with increased severity of sleep-disordered breathing

ELIGIBILITY:
Inclusion Criteria:

* Stable OSA patients

Exclusion Criteria:

* Cardiovascular diseases .
* Orthopedic or neurological conditions affecting the ability of exercise.
* Patients with previous lung resection or malignancies.
* Patients with liver cell failure, renal failure.
* Muscloskeletal disease.
* Other chronic chest disease eg, ILD.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted as prospective study including 50 patients either admitted at our chest department or presented at our out patient clinic and diagnosed as Obstructive sleep apnea according to clinical picture and sleep study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Ventilatory parameters of cardiopulmonary exercise test | 30 minutes
  End tidal Pco2 and Po2 will be measured in patients with obstructive sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Raafat T El-Sokkary, prof, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNamara SG, Grunstein RR, Sullivan CE. Obstructive sleep apnoea. Thorax. 1993 Jul;48(7):754-64. doi: 10.1136/thx.48.7.754. No abstract available. PMID 8153927
- [Background] Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004 Aug;79(8):1036-46. doi: 10.4065/79.8.1036. PMID 15301332
- [Background] Levinson PD, McGarvey ST, Carlisle CC, Eveloff SE, Herbert PN, Millman RP. Adiposity and cardiovascular risk factors in men with obstructive sleep apnea. Chest. 1993 May;103(5):1336-42. doi: 10.1378/chest.103.5.1336. PMID 8486007
- [Background] Ozturk L, Metin G, Cuhadaroglu C, Utkusavas A, Tutluoglu B. FEF(25-75)/FVC measurements and extrathoracic airway obstruction in obstructive sleep apnea patients. Sleep Breath. 2005 Mar;9(1):33-8. doi: 10.1007/s11325-005-0006-1. PMID 15785919
- [Background] Vgontzas AN, Bixler EO, Chrousos GP. Sleep apnea is a manifestation of the metabolic syndrome. Sleep Med Rev. 2005 Jun;9(3):211-24. doi: 10.1016/j.smrv.2005.01.006. PMID 15893251